CLINICAL TRIAL: NCT03692546
Title: Liposomal Bupivacaine Reduces Opiate Consumption After Rotator Cuff Repair in a Randomized Control Trial
Brief Title: Liposomal Bupivacaine for Pain Control After Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic & Neurosurgery Specialists (Other)
Responsible Party: Principal Investigator, Paul Sethi, Principal Investigator, Orthopaedic & Neurosurgery Specialists
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016017
Record Dates: First submitted 2018-09-26; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Rotator Cuff Tear; Postoperative Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (LB) (Experimental): Administration of 20 ml of LB diluted with an additional 40 ml of saline was injected into a triangular soft tissue surgical field block, along with standard bupivacaine interscalene block
  Interventions: Drug: Liposomal bupivacaine (LB)
- Interscalene Block Alone (ISB) (No Intervention): Administration of 20mL of 0.5% standard bupivacaine interscalene block with no additional soft tissue surgical field block

INTERVENTIONS:
Drug: Liposomal bupivacaine (LB) — Addition of LB solution to soft tissue surgical field block to a standard interscalene block procedure
  Other Names: EXPAREL
  Arms: Liposomal Bupivacaine (LB)

SUMMARY:
The use of an interscalene block (ISB) is often associated with rebound pain that could be avoided through adjunctive therapy with longer duration. Administration of a liposomal bupivacaine (LB) field block in addition to ISB would overcome this rebound pain to provide greater pain relief and reduce opiate consumption when compared to ISB alone. 50 patients were recruited and randomized into groups that either received or did not receive an intraoperative LB field block in addition to standard ISB administration. Visual Analog Scale (VAS) pain scores and narcotic consumption were recorded over the five-day postoperative period to determine the effectiveness of LB pain relief.

DETAILED DESCRIPTION:
Arthroscopic rotator cuff repair (ARCR) provides excellent clinical outcomes but is often associated with significant postoperative pain. As rotator cuff repair procedures become increasingly more common, these procedures and the narcotic prescriptions which accompany them may contribute to the rising opioid epidemic. The use of intraoperative local and regional anesthesia or field blocks, in conjunction with multimodal pharmacological strategies, is a widely accepted approach for managing surgical pain and reducing opiate use. The purpose of this study was to determine whether using a field block of liposomal bupivacaine (LB) in addition to an interscalene block (ISB) would provide greater pain relief and reduction in opiate consumption when compared to ISB alone.

The study enrolled 50 patients undergoing primary ARCR surgery. Patients were randomized to receiving intraoperative liposomal bupivacaine or not and provided with postoperative "Pain Journals" to document their daily pain on a visual analog scale (VAS) and to track their daily opioid consumption during the first five post-operative days.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* undergoing an arthroscopic rotator cuff repair surgery of a full thickness tear
* willing to fill out the "Pain Journal"; able to understand the informed consent process
* willing to document informed consent prior to completion of any study-related procedure
* able to read, comprehend, and complete subject-reported outcome measures in English

Exclusion Criteria:

* pregnant
* documented history of drug or alcohol abuse
* use of narcotic painkillers greater than 3 months prior to surgery
* neurologic deficit or disability involving the surgical extremity
* known allergy or intolerance to hydrocodone or oxycodone
* known allergy to amide anesthetics
* currently enrolled or planning to enroll in another clinical trial during this study that would affect the outcome of this study
* history of cognitive or mental health status that interferes with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Daily Opioid Consumption in Oral Morphine Equivalent | Post-operative day one to five
  Total amount of narcotics consumed over the study period following surgery

SECONDARY OUTCOMES:
Visual Analog Scale Pain Scores | Post-operative day one to five
  A standardized measure of subjective pain on a scale of 0 to 10, from zero pain to excruciating pain, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic & Neurosurgery Specialists, Greenwich, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber FA. Suprascapular nerve block for shoulder arthroscopy. Arthroscopy. 2005 Aug;21(8):1015. doi: 10.1016/j.arthro.2005.05.033. PMID 16086570
- [Background] Boddu C, Genza A, McCann PD. Bridging multimodal pain management provides 48-hour pain control in patients undergoing total shoulder replacement. J Shoulder Elbow Surg. 2018 Jun;27(6S):S65-S69. doi: 10.1016/j.jse.2017.12.026. Epub 2018 Feb 13. PMID 29426743
- [Background] Boss AP, Maurer T, Seiler S, Aeschbach A, Hintermann B, Strebel S. Continuous subacromial bupivacaine infusion for postoperative analgesia after open acromioplasty and rotator cuff repair: preliminary results. J Shoulder Elbow Surg. 2004 Nov-Dec;13(6):630-4. doi: 10.1016/j.jse.2004.04.005. PMID 15570231
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Chan CW, Peng PW. Suprascapular nerve block: a narrative review. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):358-73. doi: 10.1097/AAP.0b013e3182204ec0. PMID 21654552
- [Background] Chang KV, Wu WT, Hung CY, Han DS, Yang RS, Chang CH, Lin CP. Comparative Effectiveness of Suprascapular Nerve Block in the Relief of Acute Post-Operative Shoulder Pain: A Systematic Review and Meta-analysis. Pain Physician. 2016 Sep-Oct;19(7):445-56. PMID 27676661
- [Background] Ensor KL, Kwon YW, Dibeneditto MR, Zuckerman JD, Rokito AS. The rising incidence of rotator cuff repairs. J Shoulder Elbow Surg. 2013 Dec;22(12):1628-32. doi: 10.1016/j.jse.2013.01.006. Epub 2013 Mar 1. PMID 23466172
- [Background] Jacob BC, Peasah SK, Shogbon AO, Perlow ER. Postoperative Pain Management With Liposomal Bupivacaine in Patients Undergoing Orthopedic Knee and Hip Arthroplasty at a Community Hospital. Hosp Pharm. 2017 May;52(5):367-373. doi: 10.1177/0018578717715382. Epub 2017 May 1. PMID 28804154
- [Background] Kaye AD, Jones MR, Kaye AM, Ripoll JG, Galan V, Beakley BD, Calixto F, Bolden JL, Urman RD, Manchikanti L. Prescription Opioid Abuse in Chronic Pain: An Updated Review of Opioid Abuse Predictors and Strategies to Curb Opioid Abuse: Part 1. Pain Physician. 2017 Feb;20(2S):S93-S109. PMID 28226333
- [Background] Kumar K, Gulotta LV, Dines JS, Allen AA, Cheng J, Fields KG, YaDeau JT, Wu CL. Unused Opioid Pills After Outpatient Shoulder Surgeries Given Current Perioperative Prescribing Habits. Am J Sports Med. 2017 Mar;45(3):636-641. doi: 10.1177/0363546517693665. Epub 2017 Feb 9. PMID 28182507
- [Background] McLaughlin DC, Cheah JW, Aleshi P, Zhang AL, Ma CB, Feeley BT. Multimodal analgesia decreases opioid consumption after shoulder arthroplasty: a prospective cohort study. J Shoulder Elbow Surg. 2018 Apr;27(4):686-691. doi: 10.1016/j.jse.2017.11.015. Epub 2018 Jan 3. PMID 29305103
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Routman HD, Israel LR, Moor MA, Boltuch AD. Local injection of liposomal bupivacaine combined with intravenous dexamethasone reduces postoperative pain and hospital stay after shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Apr;26(4):641-647. doi: 10.1016/j.jse.2016.09.033. Epub 2016 Nov 15. PMID 27856266
- [Background] Sabesan VJ, Shahriar R, Petersen-Fitts GR, Whaley JD, Bou-Akl T, Sweet M, Milia M. A prospective randomized controlled trial to identify the optimal postoperative pain management in shoulder arthroplasty: liposomal bupivacaine versus continuous interscalene catheter. J Shoulder Elbow Surg. 2017 Oct;26(10):1810-1817. doi: 10.1016/j.jse.2017.06.044. Epub 2017 Aug 24. PMID 28844420
- [Background] Shah A, Hayes CJ, Martin BC. Characteristics of Initial Prescription Episodes and Likelihood of Long-Term Opioid Use - United States, 2006-2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 17;66(10):265-269. doi: 10.15585/mmwr.mm6610a1. PMID 28301454
- [Background] Snyder MA, Scheuerman CM, Gregg JL, Ruhnke CJ, Eten K. Improving total knee arthroplasty perioperative pain management using a periarticular injection with bupivacaine liposomal suspension. Arthroplast Today. 2016 Jan 11;2(1):37-42. doi: 10.1016/j.artd.2015.05.005. eCollection 2016 Mar. PMID 28326395
- [Background] Syed UAM, Aleem AW, Wowkanech C, Weekes D, Freedman M, Tjoumakaris F, Abboud JA, Austin LS. Neer Award 2018: the effect of preoperative education on opioid consumption in patients undergoing arthroscopic rotator cuff repair: a prospective, randomized clinical trial. J Shoulder Elbow Surg. 2018 Jun;27(6):962-967. doi: 10.1016/j.jse.2018.02.039. Epub 2018 Mar 26. PMID 29599038
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272
- [Background] Tashjian RZ, Hung M, Keener JD, Bowen RC, McAllister J, Chen W, Ebersole G, Granger EK, Chamberlain AM. Determining the minimal clinically important difference for the American Shoulder and Elbow Surgeons score, Simple Shoulder Test, and visual analog scale (VAS) measuring pain after shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Jan;26(1):144-148. doi: 10.1016/j.jse.2016.06.007. Epub 2016 Aug 18. PMID 27545048
- [Background] Tong YC, Kaye AD, Urman RD. Liposomal bupivacaine and clinical outcomes. Best Pract Res Clin Anaesthesiol. 2014 Mar;28(1):15-27. doi: 10.1016/j.bpa.2014.02.001. Epub 2014 Mar 15. PMID 24815964
- [Background] Uquillas CA, Capogna BM, Rossy WH, Mahure SA, Rokito AS. Postoperative pain control after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2016 Jul;25(7):1204-13. doi: 10.1016/j.jse.2016.01.026. Epub 2016 Apr 11. PMID 27079219
- [Background] Webb BT, Spears JR, Smith LS, Malkani AL. Periarticular injection of liposomal bupivacaine in total knee arthroplasty. Arthroplast Today. 2015 Oct 12;1(4):117-120. doi: 10.1016/j.artd.2015.09.001. eCollection 2015 Dec. PMID 28326386
- [Background] Welton KL, Kraeutler MJ, McCarty EC, Vidal AF, Bravman JT. Current pain prescribing habits for common shoulder operations: a survey of the American Shoulder and Elbow Surgeons membership. J Shoulder Elbow Surg. 2018 Jun;27(6S):S76-S81. doi: 10.1016/j.jse.2017.10.005. Epub 2017 Dec 14. PMID 29249547
- [Background] Wertheim H, Rovenstine E. Suprascapular nerve block. Anesthesiology: The Journal of the American Society of Anesthesiologists. 1941;2(5):541-545.
- [Background] Westermann RW, Anthony CA, Bedard N, Glass N, Bollier M, Hettrich CM, Wolf BR. Opioid Consumption After Rotator Cuff Repair. Arthroscopy. 2017 Aug;33(8):1467-1472. doi: 10.1016/j.arthro.2017.03.016. Epub 2017 May 29. PMID 28571723
- [Background] Yan Z, Chen Z, Ma C. Liposomal bupivacaine versus interscalene nerve block for pain control after shoulder arthroplasty: A meta-analysis. Medicine (Baltimore). 2017 Jul;96(27):e7226. doi: 10.1097/MD.0000000000007226. PMID 28682872